CLINICAL TRIAL: NCT06312696
Title: Normalizing Cervical Intersegmental Kinematics With Spinal Manipulative Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PT-2024-32814.
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Participants with chronic mechanical neck pain will be recruited and randomized into one of three groups: 1) No Treatment, 2) Light Massage (pseudo- sham), and 3) Spinal Manipulative Therapy. Using a repeated measures study design, metrics of quality of spinal motion will be compared before and after the prescribed intervention.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment group (No Intervention): No Treatment: participants will be placed in a similar position to the other groups for the same duration, but no treatment or touch will be administered.
- Pseudo sham group (Sham Comparator): Light massage group
  Interventions: Other: Light Massage
- Experimental group (Experimental): Spinal Manipulative therapy group
  Interventions: Other: SMT

INTERVENTIONS:
Other: SMT — SMT will be provided by a licensed chiropractor with at least 5 years' experience.
  Treatment will last 15 to 20 minutes each and include a brief history and examination of the cervical spine. SMT will consist of low velocity, variable amplitude spinal mobilization to the cervical spine - Maitland grades 3 or 4. Spinal segments will be determined by the chiropractor using manual palpation and the patients' response to care. Drop-table or instrument-assisted SMT will not be allowed.
  Arms: Experimental group
Other: Light Massage — Light Massage will be provided as a pseudo-sham intervention to control for time, attention, and touch by a licensed chiropractor with at least 5 years' experience to control for touch and is intended to be delivered gentler and shorter than recommended for therapeutic massage.
  Arms: Pseudo sham group

SUMMARY:
The broad long-term objective is to develop an objective biomarker for spinal health based on aberrant or abnormal movement patterns during functional activities to better target spinal manipulation therapy (SMT) and other conservative treatments. The central hypotheses are a) that aberrant spinal motions and their location (area and level) are indicative of underlying spinal dysfunction, and b) that quantified 3D cervical spine intersegmental and global motion patterns during functional tasks can be used as a biomarker for subsequent clinical studies aimed at normalizing cervical kinematics.

Specific Aim: Determine the extent to which SMT can modulate, or normalize, intersegmental motion in patients with neck pain. Rationale: SMT is a force-based biomechanical event whose hypothesized mechanism of action relies on moving the segment into the para-physiological zone, resulting in normalization of spinal kinematic function. Hypothesis: Severity of abnormal or aberrant motion, identified in those with NP, will improve following SMT. Approach: Participants with chronic mechanical neck pain will be recruited and randomized into one of three groups: 1) No Treatment, 2) Light Massage (pseudo- sham), and 3) Spinal Manipulative Therapy. Using a repeated measures study design, metrics of quality of spinal motion will be compared before and after the prescribed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific, mechanical neck pain equivalent to grades I or II (Bone and Joint Task Force on Neck Pain and Its Associated Disorders classification2 for >12 weeks
* Ages 18 to 39
* Pain intensity >3 (0-10 scale)

Exclusion Criteria:

* American Society of Anesthesiology Class III conditions and/or serious mental health conditions
* Botox injections (which resulted in clinical relief) in the past 3 months
* Chronic opioid use
* Contraindications to spinal manipulation (e.g. cervical instability; complicating neurological conditions) Spinal manipulation or mobilization of cervical spine in prior 6 months
* Ongoing non-pharmacological treatment for neck pain
* History of cervical spine surgery
* Pregnancy, currently trying to get pregnant, lactation
* Contraindications to radiation exposure

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Intersegmental and Global Range of Motion | 1 hr
  analysis will consist of calculating the percent contribution of each functional spinal unit to the overall global motion. To do that, cervical spine ROM (global and intersegmental), angular change between the beginning and end of motion, will be quantified for all planar bending directions.

SECONDARY OUTCOMES:
Neck pain intensity | 1 hr
  will be measured using the 11-box numerical rating scale (NRS). The NRS is a reliable and valid outcome measure for individuals with pain and is recommended by both the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) group and the NIH task force on research standards for back pain.
Neck disability | 1 hr
  will be measured using the Neck Disability Index (NDI), an instrument previously shown to be reliable and valid for adults with neck pain.
physical function | 1 hr
  will also be measured using the relevant domains of the PROMIS-29 Profile v2.0 Instrument - recommended by an NIH task force on research standards for back pain.
depression | 1 hr
  will also be measured using the relevant domains of the PROMIS-29 Profile v2.0 Instrument - recommended by an NIH task force on research standards for back pain.
sleep disturbance | 1 hr
  will also be measured using the relevant domains of the PROMIS-29 Profile v2.0 Instrument - recommended by an NIH task force on research standards for back pain.
Pain interference | 1 hr
  will also be measured using the relevant domains of the PROMIS-29 Profile v2.0 Instrument - recommended by an NIH task force on research standards for back pain.
Fear of pain assessment | 1 hr
  Fear-Avoidance Beliefs Questionnaire (FABQ) 68 will also be collected to assess fear of pain and aversion to physical activity/movement.
Overall function assessment | 1 hr
  The Short Form-36 (SF-36) will also be collected to assess overall function.

CONTACTS AND LOCATIONS:
Overall Officials: Arin Ellingson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States